CLINICAL TRIAL: NCT00017082
Title: A Multicenter, Phase II Study Of Oxaliplatin Single Agent As Third-Line Treatment Of Metastatic Colorectal Carcinoma
Brief Title: Oxaliplatin in Treating Patients With Recurrent Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prologue Research International (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: PROLOGUE-EFC4759; CDR0000068647 (Registry Identifier: PDQ (Physician Data Query)); SANOFI-EFC4759
Record Dates: First submitted 2001-06-06; First posted 2004-01-07 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2010-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating patients who have recurrent metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall response rate, onset and duration of partial and complete responses, and duration of stable disease in patients with recurrent metastatic colorectal cancer treated with oxaliplatin. II. Determine the overall survival of patients treated with this drug. III. Determine the proportion of patients with tumor-related symptomatic improvement and time to tumor-related symptomatic worsening in patients treated with this drug. IV. Determine the time to disease progression in patients treated with this drug. V. Determine the proportion of patients achieving stable disease when treated with this drug. VI. Determine the safety of this drug in this patient population.

OUTLINE: This is a multicenter study. Patients receive oxaliplatin IV over 120 minutes on day 1. Courses repeat every 3 weeks for up to 1 year in the absence of disease progression. Patients are followed at 30 days and then every 8 weeks for 10 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent metastatic adenocarcinoma of the colon or rectum Not amenable to potentially curative treatment (e.g., inoperable metastatic disease) Must have received 2, and only 2, prior chemotherapy regimens for metastatic or recurrent disease, including the following: First-line therapy with bolus or continuous infusion fluorouracil (5-FU) (with or without leucovorin calcium) or capecitabine OR Adjuvant therapy with 5-FU and leucovorin calcium after relapse during or within 6 months of completion of first-line therapy Second-line therapy with irinotecan or after adjuvant 5-FU and leucovorin calcium treatment failure Progressive disease by CT scan or MRI during or after first-line treatment as above OR during or within 6 months of completion of adjuvant chemotherapy as above AND during second-line irinotecan or after adjuvant treatment failure as above At least 1 unidimensionally measurable lesion At least 20 mm by CT scan or MRI At least 10 mm by spiral CT scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT and SGPT no greater than 2 times ULN (6 times ULN if liver metastases present) Alkaline phosphatase no greater than 2 times ULN (6 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No unstable angina No myocardial infarction within the past 6 months No New York Heart Association class III or IV symptomatic congestive heart failure No serious cardiac arrhythmia Pulmonary: No interstitial pneumonia or extensive and symptomatic fibrosis of the lung Other: No history of intolerance to antiemetics (e.g., 5-HT3 antagonists) or antidiarrheal medication (e.g., loperamide) to be administered concurrently with study chemotherapy No history of allergies to drugs containing platinum No known concurrent peripheral neuropathy No diabetes No active infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No other active cancer from another primary site except surgically treated non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer with an undetectable PSA level

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy, including irinotecan, for metastatic or recurrent disease and recovered No other prior first-line chemotherapy agents for metastatic or recurrent disease No prior adjuvant irinotecan No prior oxaliplatin Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy No prior radiotherapy to target lesions unless documented disease progression within the radiation portal Surgery: See Disease Characteristics More than 4 weeks since prior surgery for primary or metastatic disease and recovered Other: No prior investigational anticancer drug administered with irinotecan No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2003-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Gams, MD, Study Chair — Prologue Research International
Locations (10):
- United States (10):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Memphis Cancer Center, Memphis, Tennessee